CLINICAL TRIAL: NCT05314049
Title: Effects of Sustained Natural Apophyseal Glides (SNAGs) in Combination With McKenzie Extension Protocol (Mechanical Diagnostic Therapy) in the Management of Discogenic Low Back Pain
Brief Title: Effects of Sustained Natural Apophyseal Glides in Combination With McKenzie Extension Protocol in the Management of Discogenic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/4
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Low Back Pain; Disk Prolapse; Disk Herniated Lumbar; Sciatic Radiculopathy
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Procedure: Mckenzie Extension Protocol; Procedure: Lumbar SNAGs; Device: inferential therapy; Device: Heat Therapy
- Active Comparator Group (Active Comparator)
  Interventions: Procedure: Mckenzie Extension Protocol; Device: inferential therapy; Device: Heat Therapy

INTERVENTIONS:
Procedure: Mckenzie Extension Protocol — Mckenzie Extension Exercise Protocol will be performed by participants in prone position
Procedure: Lumbar SNAGs — Lumbar SNAGs will be performed in lumbar flexion and extension in standing Position
  Arms: Experimental Group
Device: inferential therapy — 4 pole inferential therapy in combination with superficial heating for 20 minutes
Device: Heat Therapy — superficial heating for 20 minutes

SUMMARY:
Lumbar degenerative disc disease and discogenic low back pain is comparatively common and disabling musculoskeletal condition. McKenzie's extension protocol is considered to be the gold standard physical therapy treatment for persons with acute discogenic low back pain, however the evidence is deficient in terms of additive benefits of sustained natural apophyseal glides in the management of discogenic low back pain. Thus, the current study will not only look into the positive effects of McKenzie's extension protocol in the management discogenic low back pain, but will also look into the additive benefits of sustained natural apophyseal glides in combination with McKenzie's extension protocol in the management of discogenic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants
* aged 18-50 years old
* low back pain intensity less than 80/100mm on visual analogue scale
* positive centralization phenomenon
* low signal intensity of IV disc on T2 - weighted MRI
* high intensity zone towards the posterior aspect of the disc on MRI

Exclusion Criteria:

Individuals with and any musculoskeletal, metabolic, or neurological disorders that may impair gait, postural stability or sensory integrity will be excluded from the study.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Back Pain | 2 weeks
  Pain will be measured via Visual Analogue Scale. A higher score signifies poor outcome.
Lumbar Range of Motion | 2 weeks
  Disability will be measured via inclinometer. A higher score signifies good outcome.
Postural Stability | 2 weeks
  Postural Stability will be measured via Biodex Balance System. A higher score signifies poor outcome.
Lumbar Disability | 2 weeks
  Disability will be measured via Oswestry Disability Index.

IPD SHARING:
Plan to Share IPD: No